CLINICAL TRIAL: NCT00705367
Title: A Single Center, Randomized, Placebo-Controlled, Double Blind, Parallel Group Study to Evaluate the Tolerability of a Single Dose of Abatacept 30 mg/kg Via Intravenous Infusion in Chinese SLE Subjects With Lupus Nephritis
Brief Title: Phase I Study in China - Tolerability of a Single Dose of Abatacept 30 mg/kg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM101-217
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Results first posted 2010-06-03 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Abatacept, 30 mg/kg (Active Comparator)
  Interventions: Drug: Abatacept
- Abatacept, 10 mg/kg (Other): Open-label long-term extension phase
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Placebo — Infusion, Intravenous, single dose, Day 1
  Arms: Placebo
Drug: Abatacept — Infusion, Intravenous, 30mg/kg, single dose, Day 1
  Other Names: Orencia; BMS-188667
  Arms: Abatacept, 30 mg/kg
Drug: Abatacept — Infusion, intravenous, 10 mg/kg, administered on Days 15 and 29 followed by doses every 4 weeks until the end of the study
  Other Names: Orencia; BMS-188667
  Arms: Abatacept, 10 mg/kg

SUMMARY:
The purpose of this study is to determine whether abatacept at a dose 30 mg/kg via intravenous infusion is safe and well tolerated in the treatment of lupus nephritis in mainland Chinese subjects with systemic lupus erythematosus (SLE)

ELIGIBILITY:
Inclusion Criteria:

* Men and women, at least 18 years of age, with a diagnosis of systemic lupus erythematosus (SLE) and with lupus nephritis currently stable for the last 3 months without change in treatment for lupus nephritis
* Stable renal disease
* No flaring of other organ systems in a minimum of the last 3 months

Exclusion Criteria:

* Unstable lupus nephritis and serum creatinine >3 mg/dL
* Progressive renal failure, end stage renal disease, or renal transplant requiring continuous dialysis
* Severe unstable, refractory, or progressive SLE
* History of cancer
* Participants at risk for tuberculosis
* Autoimmune disease other than SLE as main diagnosis
* Human immunodeficiency virus or herpes zoster infection
* Hepatitis-B surface antigen-positive or hepatitis C antibody-positive participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-08; Primary Completion 2009-01 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Liu MF, Wang CR, Lin LC, Wu CR. CTLA-4 gene polymorphism in promoter and exon-1 regions in Chinese patients with systemic lupus erythematosus. Lupus. 2001;10(9):647-9. doi: 10.1191/096120301682430249. PMID 11678454

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirteen (13) participants were enrolled in the short-term period of the study. Four (4/13, 30.8%) of these participants were not randomized: 3 (23.1%) no longer met study criteria after screening, and 1 (7.7%) withdrew consent. All 9 participants who completed the short-term period entered the long-term period.
Groups:
- Abatacept, 30/10 mg/kg: Short-term period: Participants received a single dose of 30-mg/kg dose of abatacept intravenously (IV) Long-term period: All participants received 10-mg/kg dose of abatacept IV on days 15 and 29 followed by doses every 4 weeks until the end of the study
- Placebo/Abatacept,10 mg/kg: Short-term period: Participants received a single dose of placebo intravenously Long-term period: Placebo arm discontinued. All participants received 10-mg/kg dose of abatacept IV on days 15 and 29 followed by doses every 4 weeks until the end of the study
Period: Short-term Period
Arm/Group | Abatacept, 30/10 mg/kg | Placebo/Abatacept,10 mg/kg
Started | 6 | 3
Completed | 6 | 3
Not Completed | 0 | 0
Period: Long-term Extension Period
Arm/Group | Abatacept, 30/10 mg/kg | Placebo/Abatacept,10 mg/kg
Started | 9 | 0
Completed | 0 | 0
Not Completed | 9 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — No longer met study criteria | 1 | 0
Not completed — Administrative reason by sponsor | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Abatacept (30 mg/kg): Infusion, Intravenous, 30 mg/kg, single dose, 24 hours
- Placebo: Infusion, Intravenous, single dose, 24 hours
- Total: Total of all reporting groups
Arm/Group | Abatacept (30 mg/kg) | Placebo | Total
Number analyzed (Participants) | 6 | 3 | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 32.50 (8.76) | 41.33 (8.33) | 35.44 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  China | 6 | 3 | 9
Duration of Lupus Nephritis [Mean (Standard Deviation); unit: months] | 41.23 (32.90) | 85.26 (65.03) | 55.90 (47.10)
Duration of Systemic Lupus Erythematosus (SLE) [Mean (Standard Deviation); unit: years] | 7.20 (5.06) | 11.11 (3.18) | 8.50 (4.73)
Weight [Mean (Standard Deviation); unit: kg] | 58.83 (10.38) | 63.67 (4.04) | 60.44 (8.79)

OUTCOME MEASURES:

1. Primary Outcome: Short-term Period: Number of Participants With Adverse Events (AEs), Serious AEs (SAEs), Deaths, Discontinuations and Infusional AEs
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. Related AE=relationship of certain, probable, possible, or missing. SAE=any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in the development of drug dependency or drug abuse, is an important medical event.
Time Frame: From Day 1 of double-blind period to 1st dose of long-term period
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Abatacept (30 mg/kg) | Placebo
Number analyzed (Participants) | 6 | 3
Participants
  Deaths | 0 | 0
  SAEs | 0 | 0
  AEs | 3 | 1
  Discontinued due to AEs | 0 | 0
  Acute infusional AEs | 0 | 0
  Peri-infusional AEs | 0 | 0

2. Secondary Outcome: Long-term Period: Number of Participants With Death as Outcome, Serious AEs (SAEs), Discontinuations Due to AEs, and Treatment-related AEs
Description: AE=any new untoward medical occurrence or worsening of a preexisting medical condition that does not necessarily have a causal relationship with this treatment. Related AE=relationship of certain, probable, possible, or missing. SAE=any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in the development of drug dependency or drug abuse, is an important medical event.
Time Frame: Days 15 to 56 days post last dose of the long-term period
Population: All participants who received at least 1 infusion of abatacept during the open-label long-term extension period of the study.
Measure: Number; unit: Participants
Groups:
- Abatacept (10 mg/kg): Long-term period: All participants received 10-mg/kg dose of abatacept IV on days 15 and 29 followed by doses every 4 weeks until the end of the study
Arm/Group | Abatacept (10 mg/kg)
Number analyzed (Participants) | 9
Participants
  Deaths | 0
  SAEs | 0
  Discontinuations due to AEs | 2
  AEs | 8
  Treatment-related AEs | 6

3. Secondary Outcome: Minimum (Cmin) Plasma Concentration of Abatacept
Description: Cmin is the minimum, or trough, concentration of a drug observed after its administration and just prior to the administration of a subsequent dose.
Time Frame: Days 15, 29, 85, 169, 253 and 337
Population: All participants who received at least 1 dose of study drug and had a serum concentration measurement relative to dosing time. n=number of evaluable participants.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Abatacept (10 mg/kg)
Number analyzed (Participants) | 9
ug/mL
  Day 15 (n=6) | 55.47 (29.356)
  Day 29 (N=9) | 42.69 (12.534)
  Day 85 (n=8) | 18.54 (11.492)
  Day 169 (n=7) | 22.66 (10.312)
  Day 253 (n=7) | 28.24 (13.883)
  Day 337 (n=4) | 25.98 (6.833)

4. Primary Outcome: Short-term Period: Number of Adverse Events (AEs) Related to Study Drug
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. Related AE=relationship of certain, probable, possible, or missing. Intensity = mild (grade 1), moderate (grade 2), severe (grade 3), life-threatening/disabling (grade 4).
Time Frame: From Day 1 of double-blind period to 1st dose of long-term period
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: Events
Arm/Group | Abatacept (30 mg/kg) | Placebo
Number analyzed (Participants) | 6 | 3
Events
  Dizziness (mild) | 1 | 0
  Oropharyngeal pain (mild) | 1 | 0
  Diarrhea (mild) | 0 | 1

5. Primary Outcome: Short-term Period: MeanSystolic and Diastolic Blood Pressure
Description: Vital sign measurements are summarized without regard to position (sitting, standing, supine).
Time Frame: Day 1 predose and postdose and Day 2
Population: All participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Abatacept (30 mg/kg) | Placebo
Number analyzed (Participants) | 6 | 3
mm Hg
  Systolic blood pressure: Day 1 predose | 129.0 (20.47) | 133.0 (8.89)
  Systolic blood pressure: Day 1 postdose | 125.8 (19.58) | 131.7 (9.29)
  Diastolic blood pressure: Day 1 predose | 84.2 (8.86) | 78.3 (12.06)
  Diastolic blood pressure: Day 1 postdose | 82.7 (9.58) | 82.7 (14.22)
  Systolic blood pressure: Day 2 | 127.5 (13.69) | 126.7 (11.55)
  Diastolic blood pressure: Day 2 | 79.5 (8.69) | 78.3 (10.41)

6. Primary Outcome: Short-term Period: Mean Heart Rate
Description: Vital signs measurements are summarized without regard to position (sitting, standing, supine).
Time Frame: Day 1 predose and postdose and Day 2
Population: All participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Abatacept (30 mg/kg) | Placebo
Number analyzed (Participants) | 6 | 3
beats per minute
  Day 1 predose | 77.0 (8.49) | 81.0 (10.15)
  Day 1 postdose | 81.2 (4.83) | 87.7 (19.60)
  Day 2 | 83.5 (4.46) | 84.0 (5.29)

7. Primary Outcome: Short-term Period: Mean Respirations Rate
Description: Vital sign measurements are summarized without regard to position (sitting, standing, supine).
Time Frame: Day 1 predose and postdose and Day 2
Population: All participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: Respirations per minute
Arm/Group | Abatacept (30 mg/kg) | Placebo
Number analyzed (Participants) | 6 | 3
Respirations per minute
  Day 1 predose | 17.7 (2.07) | 19.7 (2.08)
  Day 1 postdose | 18.7 (1.63) | 20.3 (2.52)
  Day 2 | 14.0 (3.35) | 17.3 (1.15)

8. Secondary Outcome: Maximum (Cmax) Plasma Concentration of Abatacept
Description: Cmax is a drug's maximum, or peak, concentration observed after its administration.
Time Frame: Postdosing Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Abatacept (10 mg/kg)
Number analyzed (Participants) | 4
ug/mL | 463.10 (17)

9. Primary Outcome: Short-term Period: Mean Temperature
Description: Vital sign measurements are summarized without regard to position (sitting, standing, supine).
Time Frame: Day 1 predose and postdose and Day 2
Population: All participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Abatacept (30 mg/kg) | Placebo
Number analyzed (Participants) | 6 | 3
Degrees Celsius
  Day 1 predose | 36.7 (0.51) | 36.7 (0.15)
  Day 1 postdose | 36.8 (0.59) | 36.9 (0.26)
  Day 2 | 36.9 (0.11) | 36.9 (0.12)

10. Primary Outcome: Short-term Period: Number of Participants With Clinical Laboratory and Electrocardiogram (ECG) Abnormalities
Description: Laboratory tests consisted of complete blood count, chemistry, and urinalysis.
Time Frame: Screening and Days 1 and 2
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Abatacept (30 mg/kg) | Placebo
Number analyzed (Participants) | 6 | 3
Participants
  Laboratory Abnormalities | 0 | 0
  ECG Abnormalities | 0 | 0

11. Secondary Outcome: Long-term Period: Number of Participants With Marked Abnormalities in Results of Clinical Laboratory Tests
Description: preRX=pretreatment; LLN=lower limit of normal; ULN=upper limit of normal. hemoglobin (g/dL): >3g/dL drop from preRX; hematocrit (%): <0.75*preRX; erythrocytes (*10^6 c/uL): <0.75*preRX; platelet count (*10^9 c/L): <0.67*LLN or >1.5*ULN, or <100,000/mm^3 or if preRX<LLN, use <0.5*preRX and <100,000/mm^3; leukocytes (*10^3 c/uL): <0.75*LLN, >1.25*ULN, <0.8*preRX if preRX <LLN or >1.2*preRX if preRX >ULN; >ULN if preRX <LLN, <LLN if >ULN preRX; neutrophils+bands (*10^3 c/uL): if value <1.00*10^3 c/uL; lymphocytes (*10^3 c/uL): if value <0.750*10^3 c/uL or if value >7.50*10^3 c/uL; monocytes (*10^3 c/uL): if value >2000/mm^3; basophils (*10^3 c/uL): if value >400/mm^3; eosinophils (*10^3 c/uL): if value> 0.750*10^3 c/uL
Time Frame: Days 15 to 56 days post last dose of the long-term period
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Abatacept, 30/10 mg/kg
Number analyzed (Participants) | 9
Participants
  Hemoglobin (low) | 1
  Hemoglobin (high) | NA — Not evaluated
  Hematocrit (low) | 1
  Hematocrit (high) | NA — Not evaluated
  Erythrocytes (low) | 0
  Erythrocytes (high) | NA — Not evaluated
  Platelet count (low or high) | 0
  Leukocytes (low) | 1
  Leukocytes (high) | 0
  Neutrophils +bands (absolute) (low) | NA — Not evaluated
  Neutrophils +bands (absolute) (high) | 0
  Absolute lymphocytes (low) | 6
  Absolute lymphocytes (high) | 0
  Absolute monocytes (low) | NA — Not evaluated
  Absolute monocytes (high) | 0
  Absolute basophils (low) | NA — Not evaluated
  Absolute basophils (high) | 0
  Absolute eosinophils (low) | NA — Not evaluated
  Absolute eosinophils (high) | 0

12. Secondary Outcome: Long-term Period: Number of Participants With Marked Abnormalities in Results of Clinical Laboratory Tests (Continued)
Description: preRX=pretreatment; LLN=lower limit of normal; ULN=upper limit of normal. Glucose (mg/dL): <65 or >220. Glucose, fasting(mg/dL): <0.8*LLN or >1.5* ULN; if preRX<LLN, use <0.8*preRX or >ULN; if preRX>ULN, use >2.0*preRX or <LLN. Protein, total (g/dL): <0.9*LLN or >1.1*ULN; if preRX<LLN, use 0.9*preRX or >ULN if preRX >ULN, use 1.1*preRX or <LLN. Albumin (g/dL): <0.9*LLN, or if preRX<LLN use <0.75*preRX. Uric acid (mg/dL): >1.5*ULN; if preRX>ULN use >2*preRX. Protein, urine: if missing preRX, use>=2; if >=4; if preRX=0 or 0.5, use >=2; if preRX=1, use >=3, or if preRX=2 or 3, use >= 4. Glucose, urine: if preRX missing, use >=2; if >=4, or if preRX=0 or 0.5 use >=2,or if preRX=1, use >=3, or if preRX=2 or 3 use >=4. Blood, urine: if preRX missing, use>= 2, or if >=4, or if preRX=0 or 0.5, use >=2, or if preRX=1, use >=3; if preRX=2 or 3 use >=4. WBC, urine (hpf): if missing preRX, use>= 2, or if >= 4, or if preRX =0 or 0.5 use >=2, or if preRX=1 use >=3, or if preRX=2 or 3 use >=4.
Time Frame: Days 15 to 56 days post last dose of the long-term period
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Abatacept, 30/10 mg/kg
Number analyzed (Participants) | 9
Participants
  Glucose, serum (low) | 2
  Glucose, serum (high) | 0
  Glucose, fasting serum (low) | 0
  Glucose, fasting serum (high) | 0
  Protein, total (low) | 0
  Protein, total (high) | 0
  Albumin (low) | 0
  Albumin (high) | NA — Not evaluated
  Uric acid (low) | NA — Not evaluable
  Uric acid (high) | 0
  Protein, urine (low) | NA — Not evaluated
  Protein, urine (high) | 1
  Glucose, urine (low) | NA — Not evaluated
  Glucose, urine (high) | 0
  Blood, urine (low) | NA — Not evaluated
  Blood, urine (high) | 5
  WBC, urine (low) | NA — Not evaluated
  White blood cell (WBC) count, urine (high) | 3

13. Secondary Outcome: Long-term Period: Number of Participants With Marked Abnormalities in Results of Clinical Laboratory Tests (Continued)
Description: ULN=upper limit of normal; preRX=pretreatment: ALP (U/L): >2*ULN, or if preRX>ULN, use >3*preRX; AST (U/L): >3*ULN, or if preRX>ULN, use >4*preRX; ALT (U/L): >3X*ULN, or if preRX>ULN, use >4*preRX; GGT (/L): >*ULN, or if preRX>ULN, use >3*preRX; bilirubin (mg/dL): >2*ULN, or if preRX>ULN, use >4*preRX; BUN (mg/dL):>2*preRX; sodium: <.95*LLN, >1.05*ULN, <.95* preRX if <LLN preRX, >1.05*preRX if >ULN preRX; >ULN if <LLN preRX, <LLN if >ULN preRX; potassium: chloride: calcium: phosphorous:
Time Frame: Days 15 to 56 days post last dose of the long-term period
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Abatacept, 30/10 mg/kg
Number analyzed (Participants) | 9
Participants
  Alkaline phosphatase (ALP) (low) | NA — Not evaluated
  ALP (high) | 0
  Aspartate aminotransferase (AST) (low) | NA — Not evaluated
  AST (high) | 0
  Alanine aminotransferase (ALT) (low) | NA — Not evaluated
  ALT (high) | 0
  G-glutamyl transferase (GGT) (low) | NA — Not evaluated
  GGT (high) | 0
  Bilirubin, total (low) | NA — Not evaluated
  Bilirubin, total (high) | 0
  Blood urea nitrogen (BUN) (low) | NA — Not evaluated
  BUN (high) | 0
  Sodium, serum (low) | 0
  Sodium, serum (high) | 1
  Potassium, serum (low) | 0
  Potassium, serum (high) | 0
  Chloride, serum (low) | 0
  Chloride, serum (high) | 0
  Calcium, total (low) | 0
  Calcium, total (high) | 0
  Phosphorus, inorganic (low) | 0
  Phosphorus, inorganic (high) | 2

14. Secondary Outcome: Long-term Period: Number of Participants With Abatacept-specific Antibodies
Description: Antiabatacept antibodies in human serum were assayed using a validated electrochemiluminescent immunoassay during the period of known analyte stability.
Time Frame: Day15 to 56 days post last dose of the long-term period
Population: All participants who received at least 1 dose of abatacept and had an immunogenicity test result.
Measure: Number; unit: Participants
Arm/Group | Abatacept (10 mg/kg)
Number analyzed (Participants) | 9
Participants | 0

ADVERSE EVENTS:
Arm/Group | Abatacept 30 mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 3/6 | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept 30 mg/kg (N=6) | Placebo (N=3)
DIZZINESS (Nervous system disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.